CLINICAL TRIAL: NCT01941732
Title: Motor Response to Acute Challenge to Sildenafil in Parkinsons Disease
Brief Title: Motor Response to Sildenafil in PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Winge, Consultant, ph.d., Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIA-Pilot1
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Parkinsons Disease; Erectile Dysfunction
MeSH Terms: conditions — Parkinson Disease; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental): motor function to be tested before and after challenge with 100 mg sildenafil after taking normal anti-PD medication, and Again after discontinuation of anti-PD medication for 12 h
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil
  Other Names: Sildenafil (Viagra (R)) 100 mg

SUMMARY:
Sildenafil (Viagra(R))is widely used by men with Parkinsons Disease (PD) and erectile dysfunction. A number of patients have reported that when they take Sildenafil, their need of anti-PD medication is reduced.

We hypotheses that sildenafil increases brain blood flow and hence improves the function of specific brain regions, improving motor function.

Motor function and cerebral blood flow of 8 patients will be tested before and after Sildenafil intake and before and after anti-PD medication.

DETAILED DESCRIPTION:
Erectile dysfunction can be experienced by up tp 40% of men with Parkinsons Disease (PD). Sildenafil (Viagra(R))is widely used by men with PD and erectile dysfunction. A number of patients have reported that when they take Sildenafil, their need of anti-PD medication is reduced.

We hypotheses that sildenafil increases cerebral blood flow in basal ganglia and hence improves the function, improving motor function.

Motor function and cerebral blood flow (rCBF) of 8 patients will be tested before and after Sildenafil intake and before and after anti-PD medication.

rCBF will be measured by the Xe133 inhalation method and a fast-rotating, brain-dedicated, single photon emission computerized tomograph (SPECT, Tomomatic, 232, Medimatic, Inc., Denmark). Two scans will be perfomed, when patients are i)in normal medicated state and ii) in normal medicated state 1 hour after intake of 100 mg sildenafil.

Motor function will be measured i 4 conditions: i)in normal medicated state and ii) in normal medicated state 1 hour after intake of 100 mg sildenafil, iii) after 12 hours of discontiation of anti-PD mediciation and iiii) after 14 hours of discontiation of anti-PD mediciation and 1 hour after intake of 100 mg sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Parkinsons disease
* Erectile dysfunction
* previous tried sildenafil with beneficial effects on motor function

Exclusion Criteria:

* psychosis
* Heart disease

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-11; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Motor function | 1 hour
  Motor function assessed by Unified Parkinsons disease Rating Scale, section 3 before and after challenge with Sildenafil and before and after discontinuation of anti-PD medication for 12 hours.

SECONDARY OUTCOMES:
Cerebral Blood Flow (rCBF) | 1 hour
  change in rCBF in basal ganglia from before to 1 hour after intake of 100 mg of sildenafil

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Neurology, Bispebjerg Hospital, Copenhagen, Denmark